CLINICAL TRIAL: NCT02815683
Title: Bronchoscopic Lung Volume Reduction Treatment in Clinical Practice: Introduction and Implementation in The Netherlands and Evaluation of a National Database
Brief Title: Bronchoscopic EmphysemA Treatment in THE NetherLands
Acronym: BREATHE-NL
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, MD PhD, University Medical Center Groningen
Other Study IDs: BREATHE-NL
Record Dates: First submitted 2016-06-17; First posted 2016-06-28 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: COPD
Keywords: Bronchoscopy; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: New bronchoscopic treatments for emphysema have shown promise in clinical trials, improving lung function, exercise capacity and possibly survival and are now being adopted by a number of centres in the Netherlands. It is important to ensure that the benefits seen in clinical trials are in fact reflected in clinical practice and that the best use of this early 'real world' experience is made to optimise the development and use of these novel therapies.

Overall objective: to develop a national database to record bronchoscopic lung volume reduction procedures for patients with emphysema. This is desirable for audit purposes but will also be an important resource for research both in gathering data and in facilitating collaborations.

DETAILED DESCRIPTION:
Rationale: New bronchoscopic treatments for emphysema have shown promise in clinical trials, improving lung function, exercise capacity and possibly survival and are now being adopted by a number of centres in the Netherlands. It is important to ensure that the benefits seen in clinical trials are in fact reflected in clinical practice and that the best use of this early 'real world' experience is made to optimise the development and use of these novel therapies.

Overall objective: to develop a national database to record bronchoscopic lung volume reduction procedures for patients with emphysema. This is desirable for audit purposes but will also be an important resource for research both in gathering data and in facilitating collaborations.

Study design: This study is a nationwide, multicenter, observational post-marketing study with long-term follow up (5 years).

Study population: The study population exists of patients with severe emphysema who undergo a bronchoscopic lung volume reduction treatment with one-way endobronchial valves.

Main study parameters/endpoints:

The main study parameter is the assessment of Target Lung Volume Reduction (TLVR) and correct placement of the valves at CT-scan at 30 days post treatment. This is the most accurate and directly treatment related endpoint which will also be used for quality control.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for a bronchoscopic lung volume treatment using one-way valves.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population exists of patients with severe emphysema who undergo a bronchoscopic lung volume reduction treatment with one-way endobronchial valves.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Quality of treatment | Baseline-30 days
  Quality will be assessed by a High resolution CT check at 30 day post-treatment of the placement of the valves.

SECONDARY OUTCOMES:
Change from baseline in lungfunction at 5 years follow up after treatment. | Baseline- 5 years
  -Change from baseline in lungfunction measured by the bodybox at 5 years follow up.
Change from baseline in exercise capacity at 5 years follow up after treatment. | Baseline- 5 years
  -Change from baseline in exercise capacity measured by the 6-minute walk distance test at 5 years follow up.
Change from baseline in breathlessness at 5 years follow up after treatment. | Baseline- 5 years
  -Change from baseline in breathlessness measured by the mMRC-scale (modified medical research council) at 5 years follow up.
Change from baseline in health status at 5 years follow up after treatment. | Baseline- 5 years
  -Change from baseline in health status measured by the CAT (COPD Assessment test) score at 5 years follow up.
The incidence of a pneumothorax after the treatment until 5 years follow up. | Baseline- 5 year
  The number of pneumothoraxes will be recorded between treatment and 5 years follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bakker JT, Hartman JE, Klooster K, Charbonnier JP, Tsiaousis M, Vliegenthart R, Slebos DJ. Endobronchial valve treatment improves chest-CT diaphragm configuration in COPD. Respir Med. 2024 Nov-Dec;234:107856. doi: 10.1016/j.rmed.2024.107856. Epub 2024 Nov 6. PMID 39515624
- [Derived] Hartman JE, Klooster K, Ten Hacken NHT, van Dijk M, Slebos DJ. Patient Satisfaction and Attainment of Patient-Specific Goals after Endobronchial Valve Treatment. Ann Am Thorac Soc. 2021 Jan;18(1):68-74. doi: 10.1513/AnnalsATS.202004-342OC. PMID 32881586
- See also: Website of the bronchoscopic intervention center of the UMCG — http://www.bicumcg.nl